CLINICAL TRIAL: NCT04949750
Title: Efficacy of Paper-based Cognitive Training in Vietnamese Patients With Early Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Collaborators: University of California, Davis (Other); National Geriatric Hospital (Other Government); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tống Mai Trang, Attending Physician, Neurology Department, University Medical Center, Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-VNO1002; R01AG064688 (NIH)
Record Dates: First submitted 2021-06-19; First posted 2021-07-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Early Alzheimer Disease; Paper - based cognitive training; Randomized trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper based cognitive training (Experimental): Patients with Alzheimer's disease in the early stage receive 12 weeks paper based cognitive training and standard care (medication)
  Interventions: Other: Paper - based cognitive training
- Control group (No Intervention): Patients with Alzheimer's disease in the early stage only receive standard care (medication)

INTERVENTIONS:
Other: Paper - based cognitive training — Cognitive training
  Other Names: Non pharmacological treatment for AD
  Arms: Paper based cognitive training

SUMMARY:
The purpose of this study is to assess the efficacy of paper-based cognitive training in Vietnamese patients with early Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* For patient:

  * Diagnosis of Probable Alzheimer's Disease per DSM-5 criteria;
  * In the early stage of AD (MMSE from 20 to 25);
  * Age from 60 - 80 years old;
  * Had greater than 5 years of formal education.
* For Caregiver:

  * Members (including, but not limited to partners, children, relatives, lived-in helper of the patient) that are important for care delivery and provide care-related tasks (eg personal care, eating, cooking, cleaning) and everyday decision making to the patients. They are not required to live together or spend a specific amount of time with the patients;
  * Older than 18 years of age;
  * Possess adequate Vietnamese language skills and no cognitive impairment to conduct interview and evaluation

Exclusion Criteria:

* For patient:

  * Patients with concomitant diseases (heart failure, kidney failure, liver failure or thyroid diseases) that affect cognitive functions;
  * Diagnosed with significant neurologic disease other than AD (Parkinson's disease, multi-infarct dementia, schizophrenia, history of significant head trauma followed by persistent neurologic defaults, …), major depression within the past 1 year, or taking psychoactive medications (antidepressants with significant anticholinergic side effects, neuroleptics, chronic anxiolytics or sedative hypnotics, etc) within the past 1 month;
  * Having major visual, auditory, reading, or writing impairments;
  * Patients and/or caregivers who decline to participate.
* For cargiver:

  * Having subjective complaints of cognitive impairment prevents them from understanding the instruction from the research team;
  * Having significant visual, auditory, reading, or writing impairments;
  * Caregivers who decline to participate

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Mini-Mental State Examination (MMSE) | 12 weeks from baseline cognitive assessment
  It is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. The score is between 0-30. Higher score indicating better cognition.
Change from baseline in the Memory tests | 12 weeks from baseline cognitive assessment
  Immediate Recall, Delayed Recall, Delayed Recognition are tests that measure memory function. Higher score indicating better cognition.
Change from baseline in the Trail Making test scores | 12 weeks from baseline cognitive assessment
  Raw score, assessing attention, executive function. TMT is divided into two parts, TMT-A and TMT-B. In the TMT part A, circles with number from 1 to 25 are arranged randomly. Numerical sequence should be connected by patients as quickly as possible, cutoff value > 180 seconds. In the TMT part B, patients must alternate between numbers and letters, cut off value > 300 second. Cutoff scores indicate the value above suggest cognitive performance is normal.
Change from baseline in the Digits Span forward and backward | 12 weeks from baseline cognitive assessment
  The longest digits of forward and backward are 8 and 7, respectively. The total scores are twelve for each test. Higher score indicating better cognition.
Change from baseline in the Verbal fluency test | 12 weeks from baseline cognitive assessment
  Semantic memory score will be measured using the Verbal fluency test. The verbal fluency test is a short test of verbal functioning. Participants are given 1 min to produce as many animals as possible within a semantic category (category fluency). The participant's score is the number of animals. Higher score means better cognition.
Change from baseline in the Clock drawing test | 12 weeks from baseline cognitive assessment
  1-6 points, with higher scores indicating worse visuo-spatial function.
Change from baseline in the 15-Item Version of the Boston Naming Test | 12 weeks from baseline cognitive assessment
  Cognitive test of semantic memory. Object naming to confrontation, which also depends upon intact perceptual and word retrieval ability. Higher scores indicating better cognition.
Change from baseline in the Instrumental Activities of Daily Living (IADL) score. | 12 weeks from baseline cognitive assessment
  Instrumental Activities of Daily Living (IADL) is a questionnaire to assess patient's capacity to live independently.

SECONDARY OUTCOMES:
Change from baseline in the Zarit Burden Interview (ZBI) score. | 12 weeks from baseline cognitive assessment
  Zarit Burden Interview score is a questionnaire to assess patient's caregiver burden.
Percentage of participants completes the full 12-week cognitive training. | 12 weeks from baseline cognitive assessment
  Every 4 weeks participants will follow-up at Dementia Center and be able to continue the training if they complete 80% of each level of difficulty workload. Therefore, we aim to calculate the percentage of participants who can completes the full 12-week cognitive training.

CONTACTS AND LOCATIONS:
Overall Officials: Trang M. Tong, Dr, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University Medical Center, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided